CLINICAL TRIAL: NCT02996617
Title: PEG-rhG-CSF in Patients With Non-Hodgkin Lymphoma Receiving Chemotherapy to Prevent Neutropenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wang Xin, Director of Department of Hematology, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShandongPH02
Record Dates: First submitted 2016-11-19; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma,Non-Hodgkin
Keywords: Lymphomas Non-Hodgkin's B-Cell; Lymphomas Non-Hodgkin's T-Cell; PEG-rhG-CSF; Neutropenia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, T-Cell; Neutropenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhG-CSF regimen (Active Comparator): Patients weren't preventive use of rhG-CSF（ruibai 100ug）.If their WBC≤1×10^ 9/L,they were administered rhG-CSF:5ug/kg/day until their WBC≥4×10^ 9/L for total 4 courses.
  Interventions: Drug: rhG-CSF regimen
- Pegylated rhG-CSF regimen (Experimental): Patients were administered pegylated rhG-CSF 6mg（weight≥45Kg）or 3mg（weight≤45Kg）once 24 hours after the end of chemotherapy drugs of every chemotherapy cycle for total 4 courses.
  Interventions: Drug: Pegylated rhG-CSF regimen

INTERVENTIONS:
Drug: rhG-CSF regimen — Patients weren't preventive use of rhG-CSF.If their WBC≤1×10^ 9/L,they were administered rhG-CSF:5ug/kg/day until their WBC≥4×10^ 9/L.Chemotherapy regimen: CHOP: Epirubicin：70 mg/m2 , Cyclophosphamide：750 mg/m2, Vincristine: 1.4 mg/m2 , Prednison：100mg/d; CHOPE: Epirubicin：70 mg/m2, Cyclophosphamide：750 mg/m2,Vincristine: 1.4 mg/m2,Prednison：100mg/d,Etoposide: 100 mg/（m2•d）;EPOCH:etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin;Hyper-CVAD(A):hyperfractionated cyclophosphamide, vincristine,doxorubicin, dexamethasone, cytarabine and methotrexate;GemOx-R:Gemcitabine, Oxaliplatin;GDP:gemcitabine, dexamethasone, and cisplatin
  Other Names: Pegylated rhG-CSF regimen
  Arms: rhG-CSF regimen
Drug: Pegylated rhG-CSF regimen — Patients were administered pegylated rhG-CSF 6mg（weight≥45Kg）or 3mg（weight≤45Kg）once 24 hours after the end of chemotherapy drugs of every chemotherapy cycle.Chemotherapy regimen: CHOP: Epirubicin：70 mg/m2 , Cyclophosphamide：750 mg/m2, Vincristine: 1.4 mg/m2 , Prednison：100mg/d; CHOPE: Epirubicin：70 mg/m2, Cyclophosphamide：750 mg/m2,Vincristine: 1.4 mg/m2,Prednison：100mg/d,Etoposide: 100 mg/（m2•d）;EPOCH:etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin;Hyper-CVAD(A):hyperfractionated cyclophosphamide, vincristine,doxorubicin, dexamethasone, cytarabine and methotrexate;GemOx-R:Gemcitabine, Oxaliplatin;GDP:gemcitabine, dexamethasone, and cisplatin
  Arms: Pegylated rhG-CSF regimen

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and the continuation of chemotherapy. The PEG-rhG-CSF has increased plasma half-life, and prolonged efficacy in compare with rhG-CSF. The purpose of this study is to determine the safety and effectiveness of PEG-rhG-CSF in preventing neutropenia following chemotherapy in patients with non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
Neutropenia is a common clinical complication of chemotherapy in cancer patients. It is an important factor that delays the course of standard treatments in patients. Recombinant human granulocyte colony-stimulating factor (rhG-CSF) is an effective drug for the treatment of chemotherapy-induced neutropenia. However, for patients with neutropenia, multiple rhG-CSF treatments are usually required. This is likely to extend the antitumor treatment period and increase physical and mental stress in patients. Pegylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF) is rhG-CSF chemically modified by a single methoxy polyethylene glycol group; it is able to alleviate neutropenia with a single dose. The aim of the present study was to determine the safety and effectiveness of preventive treatment with pegylated recombinant human granulocyte colony stimulating factor (PEG-rhG-CSF) on concurrent chemotherapy-induced neutropenia and to provide a rational basis for its clinical application. Therefore, the investigators designed the multi-center, open-label,randomized controlled clinical study and aimed to compare the efficacy and safety between PEG-rhG-CSF and rhG-CSF in non-Hodgkin lymphoma receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Investigator diagnosis of non-Hodgkin lymphoma(Highly invasive lymphoma/Burkitt lymphoma were excluded)
* Age 18 to 80 years
* ECOG performance status ≤ 2
* receive multi-cycle Chemotherapy naive
* grade 3/4 neutropenia occurred in the patient's first cycle chemotherapy or the risk of neutropenia >20% without rhG-CSF support
* Expected survival time≥3 months; cNormal bone marrow function(absolute neutrophil count ≥1.5 × 109/L; platelet count ≥ 80 × 109/L)
* Liver function: transaminase≤2.5× upper limit of normal value，bilirubin≤2.5×upper limit of normal value; serum creatinine≤2×upper limit of normal value;

Exclusion Criteria:

* Patients with severe complications or severe infection;
* Invasion of central nervous system;
* Patients with severe visceral organ dysfunction, heart block, myocardial infarction within 6 months;
* Prior bone marrow stem cell or organ transplantation
* patients with severe allergic constitution, or those who are allergic to Escherichia coli products; 5. Patients participate in other clinical studies within 4 weeks;
* Pregnancy, lactation
* Other patients who are not suitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3/4 neutropenia（neutrophils≤1×10^ 9/L） in every cycle | through the study completion,an average of 4 months
  Proportion of patients grade 3/4 neutropenia（neutrophils≤1×10^ 9/L）

SECONDARY OUTCOMES:
Rate of the chemotherapy delay | through the study completion,an average of 4 months
  Proportion of chemotherapy delay(>7 days) caused by neutropenia
Rate of the febrile neutropenia in every cycle | through the study completion,an average of 4 months
  Proportion of febrile caused by neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: xin wang, MD, PHD, Study Chair — Shandong Provincial Hospital
Locations (1):
- Department of Hematology, Provincial Hospital Affiliated to Shandong University, Jin'an, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Green MD, Koelbl H, Baselga J, Galid A, Guillem V, Gascon P, Siena S, Lalisang RI, Samonigg H, Clemens MR, Zani V, Liang BC, Renwick J, Piccart MJ; International Pegfilgrastim 749 Study Group. A randomized double-blind multicenter phase III study of fixed-dose single-administration pegfilgrastim versus daily filgrastim in patients receiving myelosuppressive chemotherapy. Ann Oncol. 2003 Jan;14(1):29-35. doi: 10.1093/annonc/mdg019. PMID 12488289
- [Background] Holmes FA, Jones SE, O'Shaughnessy J, Vukelja S, George T, Savin M, Richards D, Glaspy J, Meza L, Cohen G, Dhami M, Budman DR, Hackett J, Brassard M, Yang BB, Liang BC. Comparable efficacy and safety profiles of once-per-cycle pegfilgrastim and daily injection filgrastim in chemotherapy-induced neutropenia: a multicenter dose-finding study in women with breast cancer. Ann Oncol. 2002 Jun;13(6):903-9. doi: 10.1093/annonc/mdf130. PMID 12123336
- [Background] Johnston E, Crawford J, Blackwell S, Bjurstrom T, Lockbaum P, Roskos L, Yang BB, Gardner S, Miller-Messana MA, Shoemaker D, Garst J, Schwab G. Randomized, dose-escalation study of SD/01 compared with daily filgrastim in patients receiving chemotherapy. J Clin Oncol. 2000 Jul;18(13):2522-8. doi: 10.1200/JCO.2000.18.13.2522. PMID 10893282
- [Background] Hadji P, Kostev K, Schroder-Bernhardi D, Ziller V. Cost comparison of outpatient treatment with granulocyte colony-stimulating factors (G-CSF) in Germany. Int J Clin Pharmacol Ther. 2012 Apr;50(4):281-9. doi: 10.5414/cp201633. PMID 22456299
- [Background] Wen TJ, Wen YW, Chien CR, Chiang SC, Hsu WW, Shen LJ, Hsiao FY. Cost-effectiveness of granulocyte colony-stimulating factor prophylaxis in chemotherapy-induced febrile neutropenia among breast cancer and Non-Hodgkin's lymphoma patients under Taiwan's national health insurance system. J Eval Clin Pract. 2017 Apr;23(2):288-293. doi: 10.1111/jep.12597. Epub 2016 Aug 4. PMID 27491287
- [Background] Shi YK, Chen Q, Zhu YZ, He XH, Wang HQ, Jiang ZF, Chang JH, Liu YP, Wang AL, Luo DY, Zhang Y, Ke XY, Li WL, Zhang WJ, Wang XW, Zhang YP, Wang JM, Liu XQ. Pegylated filgrastim is comparable with filgrastim as support for commonly used chemotherapy regimens: a multicenter, randomized, crossover phase 3 study. Anticancer Drugs. 2013 Jul;24(6):641-7. doi: 10.1097/CAD.0b013e3283610b5d. PMID 23571496
- [Background] Molineux G. Pegylation: engineering improved pharmaceuticals for enhanced therapy. Cancer Treat Rev. 2002 Apr;28 Suppl A:13-6. doi: 10.1016/s0305-7372(02)80004-4. PMID 12173407